CLINICAL TRIAL: NCT00871299
Title: Applying Mindfulness-Based Cognitive Therapy to Treatment Resistant Depression
Brief Title: Practicing Alternative Techniques to Heal From Depression: The PATH-D Study
Acronym: PATH-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 AT004572-O1A1; R01AT004572-01A1 (NIH); 3063975; NCT01021254 (obsolete NCT alias)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Major Depressive Disorder
Keywords: Treatment-resistant depression, meditation, mindfulness
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mindfulness Based Cognitive Therapy (MBCT) + medication management
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- 2 (Active Comparator): The Health Enhancement Program (HEP) + medication management
  Interventions: Behavioral: Health Enhancement Program and medication management

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Mindfulness-Based Cognitive Therapy (MBCT) is a group treatment that integrates mindfulness meditation training with some CBT concepts and was specifically developed as a relapse prevention intervention for MDD. The program teaches skills that allow patients to disengage from habitual ("automatic") dysfunctional cognitive routines, in particular depression-related ruminative thought patterns, as a way to reduce future risk of relapse and recurrence of depression.
  Arms: 1
Behavioral: Health Enhancement Program and medication management — The Health Enhancement Program (HEP)was developed at the University of Wisconsin, Madison and is modeled after traditional activity and nutrition programs used in weight management- cardiac rehab and diabetes prevention programs. The program is designed to increase overall health and well-being by focusing on four health domains that impact health and are interventions regularly practiced at integrative medicine. These include: (I) Music Therapy (2) Nutrition (3) physical activity including, walking and stretching and (4) Functional movement.
  Arms: 2

SUMMARY:
This study is a randomized, controlled trial of Mindfulness-Based Cognitive Therapy (MBCT) versus Health-Enhancement Program (HEP) for patients with treatment-resistant major depressive disorder (MDD). Both arms of the study will continue to receive the standard medication management treatment as usual (TAU) throughout the study. MBCT is a new technique that has been found to be effective for prevention of relapse in individuals in complete recovery from depression. MBCT is a group-based, 8-week intervention that uses mindfulness meditation as its core therapeutic ingredient. It teaches people to have a different relationship to depressive thoughts and feelings. This study will use an active condition called the Health Enhancement Program (HEP) which was specifically developed to serve as a comparison condition for mindfulness interventions. HEP has been shown to decrease global stress levels and to increase perceived health. Stress has been considered a contributor to depression. One hundred and seventy four patients with MDD who have failed two or more adequate antidepressant trials will be identified and randomly assigned to one of two groups: MBCT+TAU or HEP+TAU. All patients who enroll in the study will undergo follow-up assessments at 3, 6, 9 and 12 months following the intervention. A supplemental portion of the study will enroll 88 patients to undergo functional magnetic resonance imagining (fMRI) scans immediately before and after treatment to better understand the neural pathways implicated in depression and those that may be affected through treatment.

ELIGIBILITY:
Inclusion Criteria:

DSM-IV TR Diagnosis of Major Depression receiving medication management.

Adequate trial of 2 or more antidepressants (ATHF) for a minimum of 6 weeks (one of which at UCSF).

Hamilton Depression Rating Scale 17 score ≥ 14

Any Ethnicity

English Speaking

Male or Female

No current psychotherapy (i.e. only medication management treatment) or plan to start new psychotherapy during MBCT or HEP

Exclusion Criteria:

Bipolar Disorder, Obsessive Compulsive Disorder, Schizophrenia, Schizoaffective Disorder, Antisocial and Borderline Personality Disorders, Current Eating Disorder, Pervasive Development Delay Major Depression with Psychotic Features

Active Suicidality (per HAM-D17 > 1 on item 3)

Meditation Practice once or more per week; yoga more than twice per week at study entry

Substance Abuse Disorder within 6 months

Cognitive Disorder with Mini Mental Status Exam score < 25

Medical illness rated 4 on Cumulative Illness Rating Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD-17) | Baseline, 4, 8, 24, 36, 52 week

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology(Self-Rated)-16 items(QIDS-SR16) | Baseline, weeks 1-8, 24, 36, 52 week
Short Form Health Survey-36 | Baseline, 8, 24, 36, 52 week
Clinical Global Improvement Scale (CGI) | Baseline, 8, 24, 36, 52 weeks
Work and Social Activity Scale (WSAS) | Baseline, 8, 24,36,52 weeks
Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (QLESQ-SF) | Baseline, 8, 24, 36, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Eisendrath, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Rush AJ, Trivedi M, Fava M. Depression, IV: STAR*D treatment trial for depression. Am J Psychiatry. 2003 Feb;160(2):237. doi: 10.1176/appi.ajp.160.2.237. No abstract available. PMID 12562566
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Derived] Eisendrath SJ, Gillung EP, Delucchi KL, Chartier M, Mathalon DH, Sullivan JC, Segal ZV, Feldman MD. Mindfulness-based cognitive therapy (MBCT) versus the health-enhancement program (HEP) for adults with treatment-resistant depression: a randomized control trial study protocol. BMC Complement Altern Med. 2014 Mar 11;14:95. doi: 10.1186/1472-6882-14-95. PMID 24612825
- See also: UCSF Depression Center — http://ucsfdepressioncenter.ucsf.edu/